CLINICAL TRIAL: NCT00826774
Title: Practice-based Opportunities for Weight Reduction Trial at University of Pennsylvania
Brief Title: Improving the Management of Obesity in Primary Care Practice (The Power-UP Trial)
Acronym: Power-UP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 805684; U01HL087072 (NIH)
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Obesity; Hypercholesterolemia; Metabolic Syndrome; Hypertension; Diabetes
Keywords: Body Weight; Overweight; Hypertension; Hyperglycemia
MeSH Terms: conditions — Obesity; Hypercholesterolemia; Metabolic Syndrome; Hypertension; Diabetes Mellitus; Body Weight; Overweight; Hyperglycemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ususal Care (Active Comparator)
  Interventions: Behavioral: Usual Care
- Breif Lifestyle Counseling (Experimental)
  Interventions: Behavioral: Brief Lifestyle Counseling
- Enhanced Brief Lifestyle Counseling (Experimental)
  Interventions: Behavioral: Enhanced Brief Lifestyle Counseling

INTERVENTIONS:
Behavioral: Usual Care — Participants in this group will receive usual medical care, provided by their own primary care providers (PCPs). PCPs also will provide participants recommendations for weight management at quarterly-scheduled visits.
  Arms: Ususal Care
Behavioral: Brief Lifestyle Counseling — These participants, like those in the Usual Care group, will receive the same PCP visits, plus monthly brief counseling sessions with an auxiliary health care provider (e.g., a medical assistant), on-site or by phone.
  Arms: Breif Lifestyle Counseling
Behavioral: Enhanced Brief Lifestyle Counseling — These participants will receive the same intervention as those in the Brief Lifestyle Counseling condition, including quarterly PCP visits and monthly sessions with a medical assistant who will instruct them in lifestyle modification. These individuals also will select, in consultation with their PCP, the use of either meal replacements or weight loss medication, to facilitate the induction and maintenance of weight loss
  Arms: Enhanced Brief Lifestyle Counseling

SUMMARY:
The purpose of the study is to compare three methods of achieving weight loss in primary care medical practice. The study will be conducted in six primary care practices. Weight management will be provided to a total of 390 obese patients (who have 2 or more components of the metabolic syndrome) by their own primary care providers, in conjunction with the practices' auxiliary health professionals, including medical assistants.

DETAILED DESCRIPTION:
Obesity, defined by a body mass index (BMI) ≥ 30 kg/m2, affects more than 31% of American adults. Additionally, nearly one-quarter of U.S. adults meet criteria for the metabolic syndrome, a clustering of clinical signs (i.e., elevated waist circumference, blood pressure, glucose or triglycerides, decreased HDL cholesterol) that is associated with increased risk of cardiovascular death. Behavior modification programs and pharmacologic interventions for obesity typically result in an 8% to 10% loss of initial body weight. Losses of this magnitude are associated with clinically significant improvements in metabolic parameters among obese persons. The availability of traditional behavioral weight control programs, however, is limited as many of these programs are based in academic medical centers. Furthermore, pharmacotherapy is seldom covered by third-party payers. Thus, there are concerns about the accessibility of these interventions to the many obese individuals who could benefit from weight loss.

The purpose of the study is to improve the management of obesity in primary care practice, where obesity is commonly encountered but infrequently addressed. Three hundred and ninety persons at 6 primary care practices within the University of Pennsylvania Health System will be randomized to one of three 2-year interventions: Usual Care, Brief Lifestyle Counseling, or Enhanced Brief Lifestyle Counseling. After training in obesity management and intervention strategies, each site will enroll approximately 65 individuals with a BMI of 30-50 kg/m2 plus two or more components of the metabolic syndrome. Participants in the Usual Care condition (N=130) will receive educational materials plus quarterly visits with a primary care provider (PCP). Those in the Brief Lifestyle Counseling condition (N=130) will receive the same PCP visits, plus 26 brief counseling sessions with an auxiliary health care provider (e.g., a medical assistant), on-site or by phone. Participants in the Enhanced Brief Lifestyle Counseling condition (N=130) will additionally receive the same treatment as those in the Brief Lifestyle Counseling group, plus the choice of adjunctive meal replacements or pharmacotherapy.

Two-year changes in weight will be compared across groups. Participants who receive the Brief Lifestyle Counseling and the Enhanced Brief Lifestyle Counseling interventions are predicted to achieve greater weight loss than those who receive Usual Care. A secondary hypothesis is that participants in Enhanced Brief Lifestyle Counseling condition will lose significantly more weight at month 24 than participants in the Brief Lifestyle Counseling group. Secondary analysis will also compare changes in the metabolic syndrome (and its individual components), mood, quality of life, dietary intake, eating behavior, appetite, physical activity and sexual function, as well as cost-effectiveness, among the three conditions. Intervention protocols and study results will be disseminated to other health care providers and payers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years

  * BMI 30-50 kg/m2 and weight ≤ 400 lbs.
  * At least 2 of 5 criteria for metabolic syndrome

    * Elevated waist circumference (> 102 cm for men, > 88 cm for women)
    * Elevated blood pressure (≥ 130/85 mmHg)
    * Impaired fasting glucose (≥ 100 mg/dl)
    * Elevated triglycerides (≥ 150 mg/dl)
    * Low HDL cholesterol (< 40 for men, < 50 mg/dl for women)
  * Willing to change diet, physical activity and weight
  * Willing to accept randomization to each group
  * Able to give informed consent
  * Patient of participating PCP

Persons with the following conditions are eligible with PCP approval:

* Diabetes mellitus
* Prior CVD event > 6 months before randomization
* Stable CVD or peripheral vascular disease

Exclusion Criteria:

* Serious medical condition likely to hinder accurate measurement of weight, or for which weight loss is contraindicated, or which would cause weight loss (e.g., end-stage renal disease on dialysis, cancer diagnosis or treatment within 2 yrs)
* Prior or planned bariatric surgery
* Chronic use (at least past 6 months) of medications likely to cause weight gain or prevent weight loss (e.g. corticosteroids, lithium, olanzapine, risperidone, clozapine)
* Unintentional weight loss within 6 months of enrollment (≥ 5% of body weight)
* Intentional weight loss within 6 months of enrollment (≥ 5% of body weight)
* Pregnant or nursing within past 6 months
* Plans to relocate from the area within 2 years
* Another member of household is a study participant or staff in the trial
* Consumes > 14 alcoholic drinks per week
* Current use of illicit substances
* Psychiatric hospitalization in last year
* Psychiatric condition likely to impair adherence to treatment (e.g., schizophrenia)
* Blood pressure ≥ 160/100 mmHg; patient may be re-screened in 1 month
* Principal Investigator or PCP discretion

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2008-01; Primary Completion 2011-02 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Weight | Measured at Month 24

SECONDARY OUTCOMES:
Prevalence of the metabolic syndrome | at 24 months
Blood Pressure | at 24 months
Lipid levels | at 24 months
Sexual function | at 24 months
Mood | at 24 months
Homeostasis model assessment of insulin resistance (HOMA-IR) | at 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Wadden, PhD, Principal Investigator — University of Pennsylvania

REFERENCES:
- [Derived] Wadden TA, Volger S, Sarwer DB, Vetter ML, Tsai AG, Berkowitz RI, Kumanyika S, Schmitz KH, Diewald LK, Barg R, Chittams J, Moore RH. A two-year randomized trial of obesity treatment in primary care practice. N Engl J Med. 2011 Nov 24;365(21):1969-79. doi: 10.1056/NEJMoa1109220. Epub 2011 Nov 14. PMID 22082239
- [Derived] Yeh HC, Clark JM, Emmons KE, Moore RH, Bennett GG, Warner ET, Sarwer DB, Jerome GJ, Miller ER, Volger S, Louis TA, Wells B, Wadden TA, Colditz GA, Appel LJ. Independent but coordinated trials: insights from the practice-based Opportunities for Weight Reduction Trials Collaborative Research Group. Clin Trials. 2010 Aug;7(4):322-32. doi: 10.1177/1740774510374213. Epub 2010 Jun 23. PMID 20573639